CLINICAL TRIAL: NCT03560193
Title: An Open Label, Multicenter, Randomized Trial of 2% Chlorhexidine-70% Isopropanol vs 5% Povidone Iodine-69% Ethanol for Skin Antisepsis in Reducing Surgical-site Infection After Cardiac Surgery
Brief Title: Randomized Trial of 2% Chlorhexidine-70% Isopropanol vs 5% Povidone Iodine-69% Ethanol for Skin Antisepsis in Reducing Surgical-site Infection After Cardiac Surgery
Acronym: CLEAN2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CLEAN2
Record Dates: First submitted 2018-05-24; First posted 2018-06-18 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Cardiac Surgery in Adult Patient
Keywords: Skin antisepsis; Chlorhexidine; Povidone Iodine; Surgical site infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chlorhexidine Group (Experimental)
  Interventions: Drug: 2%Chlorhexidine-70%Isopropanol
- Povidone Iodine Group (Active Comparator)
  Interventions: Drug: 5%Povidone Iodine- 69%Ethanol

INTERVENTIONS:
Drug: 2%Chlorhexidine-70%Isopropanol — 2% Chlorhexidine-70% isopropanol will be used to disinfect the skin before Cardiac Surgery and during all dressing changes
  Arms: Chlorhexidine Group
Drug: 5%Povidone Iodine- 69%Ethanol — 5%Povidone Iodine- 69%Ethanol will be used to disinfect the skin before Cardiac Surgery and during all dressing changes
  Arms: Povidone Iodine Group

SUMMARY:
Despite completion of more than 9 million procedures each year in France, the best antiseptic solution to be used for preparing the skin to reduce risk of surgical site infection (SSI) remains unknown. 2% Chlorhexidine gluconate (CHG)-alcohol is superior to Povidone Iodine (PVI)-alcohol for short term vascular catheter care (Mimoz O, Lancet 2015; Pages J, Intensive Care Med 2016), but studies comparing both antiseptic solutions for clean-contaminated surgical procedures led to conflicting results.

The present study will be the first large scale multicenter randomized controlled trial adequately powered to compare efficacy and safety of CHG-alcohol over PVI-alcohol in reducing SSI after clean surgery.

A clean surgery was chosen because pathogens involved in SSI mostly originate from skin. Therefore, optimisation of skin disinfection before surgery has the potential to reduce the incidence of SSI. Cardiac surgery was chosen because SSI may be severe, diagnosis of SSI is easy to monitor and to define and infections arise earlier than other frequent clean surgeries using implants such as orthopaedic or vascular surgery.

The incidence of reoperation for any purpose will be used as the main objective because there are easy to track and define and are less susceptible to interpretation in an open trial than superficial SSI. According to CDC criteria, patients will be monitored up to Day 90 because mediastinitis after cardiac surgery may occur after the usual 30-day SSI surveillance period.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥ 18 years)
* Undergoing any (scheduled) surgery of the heart (valve, coronary or combined surgery) or of the aorta via a median sternotomy
* Having given their informed consent

Exclusion Criteria:

* Patients with known allergies to CHG, PVI, isopropanol or ethanol
* Surgery for heart transplantation
* Any signs of inflammation or sternal instability at the site of sternotomy or operation for infection (SWI or endocarditis)
* Patients with history of cardiac surgery within 3 months preceding enrolment
* Participation to another clinical trial aimed at reducing SSI
* Patients already enrolled in this study
* Pregnant or breastfeeding women
* Women at age to procreate and not using effective contraception
* Patients not benefiting from a Social Security scheme or not benefiting from it through a third party
* Persons benefiting from enhanced protection, namely minors, persons deprived of their liberty by a judicial or administrative decision, adults under legal protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3316 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Incidence of any re-sternotomy occurring between Day 0 and Day 90 after surgery | 90 days
Incidence of any reoperation on saphen venous/radial artery site occurring between Day 0 and Day 30 after surgery. | 30 days

SECONDARY OUTCOMES:
Incidence of mediastinitis according to CDC criteria occurring by Day 90 after surgery and pathogens involved | 90 days
Incidence of deep incisional SSIs at saphen venous/radial artery site according to CDC criteria occurring by Day 30 after surgery and pathogens involved | 30 days
Incidence of superficial incisional SSIs at sternal or saphen venous/radial artery sites according to CDC criteria occurring by Day 30 after surgery and pathogens involved | 30 days
Incidence of SWI requiring reoperation, occurring by Day 90 | 90 days
Incidence of SSIs at saphen venous/radial artery site requiring reoperation, occurring by Day 30 | 30 days
Incidence of unexpected need for re-admission to the ICU or re-hospitalisation | 90 days
Number of days in ICU | 90 days
Number of days under mechanical ventilation | 90 days
Number of days in Hospital | 90 days
Number of days in rehabilitation unit | 90 days
Mortality at Day 90 of surgery | 90 days
Incidence of local and systemic side effects possibly linked to antiseptic use | 90 days
Economic analysis including cost-effectiveness of surgical skin antisepsis | 90 days

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - University Hospital of Clermont-Ferrand, Clermont-Ferrand
  - University Hospital of Nantes, Nantes
  - La Pitié Salpétrière Hospital, Paris
  - Institut Mutualiste Montsouris, Paris
  - University Hospital of Poitiers, Poitiers
  - University Hospital of Rennes, Rennes
  - CHRU de Strasbourg, Strasbourg
  - CHU de Toulouse, Toulouse

REFERENCES:
- [Derived] Boisson M, Corbi P, Kerforne T, Camilleri L, Debauchez M, Demondion P, Eljezi V, Flecher E, Lepelletier D, Leprince P, Nesseler N, Nizou JY, Roussel JC, Rozec B, Ruckly S, Lucet JC, Timsit JF, Mimoz O. Multicentre, open-label, randomised, controlled clinical trial comparing 2% chlorhexidine-70% isopropanol and 5% povidone iodine-69% ethanol for skin antisepsis in reducing surgical-site infection after cardiac surgery: the CLEAN 2 study protocol. BMJ Open. 2019 Jun 17;9(6):e026929. doi: 10.1136/bmjopen-2018-026929. PMID 31213447